CLINICAL TRIAL: NCT02243748
Title: Translation of a Lung Cancer Palliative Care Intervention for Clinical Practice
Brief Title: Palliative Care Intervention in Improving Symptom Control and Quality of Life in Patients With Stage II-IV Non-small Cell Lung Cancer and Their Family Caregivers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 14206; NCI-2014-01926 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 14206 (Other: City of Hope Medical Center); 1R01NR015341-01 (NIH)
Record Dates: First submitted 2014-09-16; First posted 2014-09-18 (Estimated); Last update posted 2019-05-08 (Actual); Status verified 2019-05

CONDITIONS: Caregiver; Psychological Impact of Cancer and Its Treatment; Recurrent Non-small Cell Lung Cancer; Stage IIA Non-small Cell Lung Cancer; Stage IIB Non-small Cell Lung Cancer; Stage IIIA Non-small Cell Lung Cancer; Stage IIIB Non-small Cell Lung Cancer; Stage IV Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Palliative Care; Patient Comfort

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Phase I (usual care) (Active Comparator): Participants receive usual care. This phase will aid in identifying usual care patterns in each site and provide an audit of system utilization as well as finalization of the educational materials for Phase II.
  Interventions: Other: quality-of-life assessment; Other: questionnaire administration
- Phase II (individualized palliative care) (Experimental): Participants receive individualized palliative care comprised of tailored educational sessions designed for each patient and FCG that have been modified based on patterns observed in Phase I. The first patient teaching session will cover physical and psychological areas and the second will cover social and spiritual areas. These sessions will be completed within 2 weeks of accrual. A third teaching session is held with the FCG alone to give the FCG the opportunity to discuss their perspectives and focus on their needs. Patients will be asked to identify topics they want included and which if any should be omitted which provides for tailoring of the content to the patient's needs and preferences.
  Interventions: Other: Palliative Therapy; Other: quality-of-life assessment; Other: questionnaire administration

INTERVENTIONS:
Other: Palliative Therapy — Receive individualized palliative care
  Other Names: Comfort Care; Palliative Care; Palliative Treatment; Symptom Management
  Arms: Phase II (individualized palliative care)
Other: quality-of-life assessment — Ancillary studies
  Other Names: quality of life assessment
Other: questionnaire administration — Ancillary studies

SUMMARY:
This clinical trial studies a palliative care intervention in improving symptom control and quality of life in patients with stage II-IV non-small cell lung cancer and their family caregivers. Palliative care programs can provide patients and their caregivers with information on how to manage their symptoms, maintain health and well-being, and access supportive care services. An interdisciplinary palliative care model may effectively link lung cancer patients to the appropriate supportive care services in a timely fashion.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Adapt a Palliative Care Intervention (PCI) tested in a National Cancer Institute (NCI) funded Program Project (P01) for dissemination to other oncology settings.

II. Determine the impact of the PCI on patient outcomes including symptom control, quality of life (QOL), and distress as compared to the usual care group.

III. Determine the impact of the PCI on family caregivers (FCG) outcomes including caregiver burden, caregiver distress, skills preparation and QOL as compared to the usual care group.

IV. Test the effects of the PCI on patient resource utilization as compared to the usual care group.

OUTLINE: Participants are enrolled sequentially to 1 of 2 phases.

PHASE I: Participants receive usual care. This phase will aid in identifying usual care patterns in each site and provide an audit of system utilization as well as finalization of the educational materials for Phase II.

PHASE II: Participants receive individualized palliative care comprised of tailored educational sessions designed for each patient and FCG that have been modified based on patterns observed in Phase I. The first patient teaching session will cover physical and psychological areas and the second will cover social and spiritual areas. These sessions will be completed within 2 weeks of accrual. A third teaching session is held with the FCG alone to give the FCG the opportunity to discuss their perspectives and focus on their needs. Patients will be asked to identify topics they want included and which if any should be omitted which provides for tailoring of the content to the patient's needs and preferences.

In both groups, participants are followed up for 3 months.

ELIGIBILITY:
Inclusion Criteria:

Patient eligibility criteria for entry into the project include:

* Diagnosis of stages II-IV non-small cell lung cancer (NSCLC)
* Undergoing treatment with surgery, chemotherapy, radiation, or combined modalities
* In Phase 2, subjects are also required on accrual to be referred to Palliative Care

FCG eligibility criteria include:

* Designated by the patient as a person closely involved in their care
* Age 18 years and older

All subjects must have the ability to understand and the willingness to sign a written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 361 (Actual)
Dates: Start 2015-02; Primary Completion 2019-04 (Actual); Study Completion 2019-04-22 (Actual)

PRIMARY OUTCOMES:
Impact of the PCI on symptom control as compared to the usual care group | Up to 3 months
  The demographic and clinical characteristics as well as baseline symptom control scores in the two phases will be compared. A repeated measures mixed model will be utilized for the three repeated measures (0, 1, and 3 months).
Impact of the PCI on patient QOL as compared to the usual care group | Up to 3 months
  The demographic and clinical characteristics as well as baseline QOL scores in the two phases will be compared. A repeated measures mixed model will be utilized for the three repeated measures (0, 1, and 3 months).
Impact of the PCI on psychological distress as compared to the usual care group | Up to 3 months
  The demographic and clinical characteristics as well as baseline psychological distress scores in the two phases will be compared. A repeated measures mixed model will be utilized for the three repeated measures (0, 1, and 3 months).
Impact of the PCI on caregiver burden as compared to the usual care group | Up to 3 months
  The demographic and clinical characteristics as well as baseline caregiver burden scores in the two phases will be compared. A repeated measures mixed model will be utilized for the three repeated measures (0, 1, and 3 months).
Impact of the PCI on caregiver distress as compared to the usual care group | Up to 3 months
  The demographic and clinical characteristics as well as baseline caregiver distress scores in the two phases will be compared. A repeated measures mixed model will be utilized for the three repeated measures (0, 1, and 3 months).
Impact of the PCI on caregiver skills preparation as compared to the usual care group | Up to 3 months
  The demographic and clinical characteristics as well as baseline caregiver skills preparation scores in the two phases will be compared. A repeated measures mixed model will be utilized for the three repeated measures (0, 1, and 3 months).
Impact of the PCI on caregiver QOL as compared to the usual care group | Up to 3 months
  The demographic and clinical characteristics as well as baseline caregiver QOL scores in the two phases will be compared. A repeated measures mixed model will be utilized for the three repeated measures (0, 1, and 3 months).
Effects of the PCI on resource utilization as compared to the usual care group | Up to 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Betty Ferrell, Principal Investigator — City of Hope Medical Center; Huong Nguyen, MD, Principal Investigator — Kaiser Permanente Department of Research and Evaluation
Locations (5):
- United States (5):
  - City of Hope Medical Center, Duarte, California
  - Southern California Permanente Medical Group, Irvine, California
  - Kaiser Permanente-Ontario Vineyard Medical Offices and Ambulatory SurgiCenter, Ontario, California
  - Kaiser Permanente Department of Research and Evaluation, Pasadena, California
  - Kaiser Permanente Medical Center, Riverside, California

REFERENCES:
- [Derived] Nguyen HQ, Cuyegkeng T, Phung TO, Jahn K, Borneman T, Macias M, Ruel N, Ferrell BR. Integration of a Palliative Care Intervention into Community Practice for Lung Cancer: A Study Protocol and Lessons Learned with Implementation. J Palliat Med. 2017 Dec;20(12):1327-1337. doi: 10.1089/jpm.2017.0143. Epub 2017 Jun 9. PMID 28598227